CLINICAL TRIAL: NCT05700630
Title: MT2022-06: Phase I Study of FT538 Monotherapy and in Combination With Vorinostat for the Treatment of Persistent Low-Level HIV Viremia
Brief Title: Ph1 Study of FT538 Alone and With Vorinostat for Persistent Low-Level HIV Viremia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Abandoned
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2022LS028
Record Dates: First submitted 2022-12-09; First posted 2023-01-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: HIV-1-infection; ART; Cd4+ Lymphocyte Deficiency; Lymphoid Tissue; Infection; Interleukin
Keywords: FT538; ACC/AHA; ADCC; AE; AIDS; ASCVD; CAR; CFR; CIBMTR; CLIA; CNS; CRP; CRS; CSRC; DC; DLT; GALT; HDACi; HIV; ICANS; ICE; IL-15; pVL
MeSH Terms: conditions — Cd4+ Lymphocyte Deficiency; Infections; Acquired Immunodeficiency Syndrome | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Determine the safety and feasibility of administering FT538 monotherapy (Experimental): Administering FT538 monotherapy as an intravenous infusion once every 14 days for 4 consecutive doses and in combination with twice weekly vorinostat for the reduction of the HIV reservoir.
  Interventions: Biological: FT538
- Characterize the toxicities and impact of FT538 and vorinostat (Experimental): To characterize the toxicities associated with FT538 monotherapy and with vorinostat in this patient population. To determine the impact of FT538 on the persistence of low-level HIV viremia, defined as detectable HIV-1 RNA of ≤200 copies/mL despite good ART adherence.
  Interventions: Biological: FT538; Drug: Vorinostat

INTERVENTIONS:
Biological: FT538 — FT538 is an investigational off-the-shelf cryopreserved NK cell product derived from an iPSC that contains three functional modifications: 1) a novel high affinity, non-cleavable CD16 (Fc receptor) that maintains CD16 on the cell surface and remains fully functional after NK cell activation, thus augmenting ADCC; 2) an IL-15 receptor fusion that promotes NK cell activity and enhances cell persistence; and 3) the knock-out of CD38 expression prevent anti-CD38 antibody-induced fratricide.
Drug: Vorinostat — Vorinostat is a histone deacetylase inhibitor (HDACi) that is FDA approved for the treatment of cutaneous T-cell lymphoma and, under investigation in HIV as disruptor of HIV latency.
  Arms: Characterize the toxicities and impact of FT538 and vorinostat

SUMMARY:
This is a single center Phase I clinical trial of FT538 administered intravenously (IV) once every 14 days for 4 consecutive doses for the reduction of the HIV reservoir in lymphoid tissue of HIV-infected individuals receiving standard of care (SOC) antiretroviral therapy (ART). As this is an early 1st in human study and the 1st for HIV-infected individual, the safety of FT538 is confirmed prior to the addition of oral vorinostat to explore the concept of "Kick and Kill".

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥18 and ≤65 years at the time of signing the consent form
* HIV-1 infection on continuous antiretroviral therapy (ART) for at least 12 months without any interruptions of greater than 14 consecutive days and without plans to modify ART before the End of Treatment visit.
* Two or more consecutive detectable HIV RNA levels of ≤200 copies/mL in the last 2 years, with at least one determination meeting this criterion in the previous 12 months. (If testing was not obtained within 42 days of planned dose 1, test will be repeated during subject screening to confirm status)
* Screening CD4+ T cell count ≥350 cells/ µl within 28 days of the 1st dose of FT538.
* Completion of initial COVID-19 vaccination series and/or documented COVID-19 infection with completion of treatment ≥ 3 months prior
* Patient weight of ≥ 50 kg due to FT538 fixed cell dosing and FT538 product pre-dosed packaging.

Adequate organ function within 14 days of Day 1, defined as the following:

* Platelet counts >150,000/mm^3
* Hemoglobin > 12.5 g/dL for men and > 11.5 g/dL for women. It is not acceptable for patients to be transfused within the prior month to meet this requirement. The use of Epogen is permitted.
* AST and ALT ≤ 3 x upper limit of institutional normal
* Estimated CrCl (eGFR) >50 mL/min/1.73m^2
* Persons of childbearing potential or with partners of childbearing potential must be willing to abstain from heterosexual activity or to use a highly effective form of contraception from the time of study enrollment through at least 4 months after the last dose of FT538. Persons are considered of childbearing potential unless: they are postmenopausal; are surgically sterile; or they have a congenital or acquired condition that prevents childbearing. NOTE: Abstinence is acceptable if this is the usual lifestyle and preferred contraception.

For Dose Cohort 4 (FT538 plus Vorinostat):

* Females of childbearing potential must use highly effective contraception from the time of study enrollment through 6 months after the last dose of vorinostat.
* Males with partners of childbearing potential must use highly effective contraception from the time of study enrollment through 3 months after the last dose of vorinostat or 4 months after the last dose of FT538, whichever is more conservative.
* Must agree to and sign the consent for the Master Long-Term Follow-Up study to fulfill the FDA recommended 15 years following exposure to the investigational gene therapy product.
* Voluntary written consent prior to the performance of any research related procedures.

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control for a minimum of 4 months after the last dose of FT538. If of childbearing potential, a negative pregnancy test is required within 14 days prior to the 1st dose of FT538 or within 7 days prior to the 1st dose of vorinostat if treated in Dose Cohort 4.
* Known allergy to the following FT538 components: albumin (human) or DMSO.
* Currently receiving or likely to require systemic immunosuppressive therapy (e.g., prednisone >5 mg daily) for any reason within 5 days before the 1st dose of FT538 and 14 days after the last dose of FT538 - inhaled and topical steroids are permitted.
* Active or recent malignancy requiring systemic chemotherapy or surgery in the preceding 36 months or for whom such therapies are expected in the subsequent 12 months - minor surgical removal of localized skin cancers (squamous cell carcinoma, basal cell carcinoma) is permitted.
* Prior history of solid organ transplant or hematopoietic stem cell transplant.
* Receipt of any investigational agent (not approved by the FDA for any indication) within 28 days prior to the first dose of FT538. Note that participation in prior HIV cure studies, including those involving IL-2 or N803, is permitted as long as experimental therapy completed >28 days prior.
* Chronic liver disease defined as Class B and C on the Child-Pugh scale.
* Active and poorly controlled atherosclerotic cardiovascular disease (ASCVD), as defined by 2013 ACC/AHA guidelines, including a previous diagnosis of any of the following within the previous 12 months: (a) acute myocardial infarction, (b) acute coronary syndromes, (c) stable or unstable angina, (d) coronary or other arterial revascularization, (e) stroke, (f) transient ischemic attack (TIA), or (g) peripheral arterial disease presumed to be of atherosclerotic origin.
* Moderate-severe obstructive lung disease. In subjects reporting a history of mild obstructive lung disease at screening, pulmonary function test (PFT) to be obtained and patient excluded from study if the FEV1 is <80% of predicted.
* Non-malignant CNS disease such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease or receipt of medications for these conditions in the 2-year period leading up to study enrollment.
* Known concurrent or recent (defined as having received treatment within the last 3 months) infection with:

  * Latent or active TB infection prior to completing a standard regimen of anti-TB therapy; defined as meeting PPD criteria for TB exposure or a positive quantiferon gold test collected at screening
  * Active fungal infection requiring systemic antifungal therapy
  * Chronic active hepatitis B or C. For Hepatitis B this will be defined as HBs antigen + and for Hepatitis C this will be defined as Hepatitis C antibody positive and Hepatitis C PCR+.
  * COVID-19; defined as a positive SARS-CoV-2 PCR test at screening or a history of COVID-19 diagnosed within the last 3 months.
* Clinical vaccination administered within 6 weeks of the 1st dose of FT538.
* Presence of any social issues that, per investigator judgement, are likely to interfere with study conduct or may cause increased risk to patient.
* Patient history of alcohol or substance abuse that, per investigator judgement, are likely to interfere with study conduct or may cause increased risk to patient
* Any medical condition or clinical laboratory abnormality that, per investigator judgement, precludes safe participation in and completion of the study or that could affect compliance with protocol conduct or interpretation of results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2024-07-26 (Estimated); Study Completion 2024-08-21 (Estimated)

PRIMARY OUTCOMES:
Determine the safety and feasibility of administering FT538 monotherapy. | 26 months
  At screen and baseline visits, all grades of signs and symptoms that occurred 30 days prior to the visit will be recorded. At all subsequent visits, all grades of signs and symptoms that occurred since the previous visit must be recorded as part of an Adverse Event (AE) assessment.

SECONDARY OUTCOMES:
Characterize the toxicities associated with FT538 monotherapy and vorinostat. | 30 months
  flow cytometric analysis for NK cell degranulation (CD107a).
Determine the impact of FT538 on the persistence of low-level HIV viremia | 30 months
  Defined as patients with detectable HIV-1 RNA of ≤200 copies/mL despite good ART adherence.

OTHER OUTCOMES:
Characterize FT538 and Vorinostat Relationship with HIV RNA | 30 months
  Ultrasensitive qPCR diagnostics will be used to quantify ratio of HIV RNA to single-copy levels.
FT538 impact on frequency and phenotype of viral cells in PBMC lymphocyte subsets. | 30 months
  Detection of viral antigens using an ultra-sensitive p24 system.
Optional lymphoid tissue collection | 30 months
  To determine the impact of FT538 on the frequency, location, and phenotype of viral RNA-positive and DNA-positive cells in lymphoid tissues (inguinal lymph node and colonic)

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Research related samples will be managed using established protocols in the Schacker Laboratory.